CLINICAL TRIAL: NCT07055919
Title: A Prospective, Multicenter, Stratified Randomized Controlled, Non-Inferiority Clinical Trial to Evaluate the Safety and Efficacy of the Structural Heart Surgery Assist System for Transcatheter Mitral Valve Edge-to-Edge Repair (TEER).
Brief Title: Structural Heart Surgery Assist System for Transcatheter Mitral Valve Edge-to-Edge Repair (TEER).
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiamen Cardiovascular Hospital, Xiamen University (Other)
Responsible Party: Principal Investigator, Yan Wang, Principal Investigator, Xiamen Cardiovascular Hospital, Xiamen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QX2025-001-02; Beijing Jiekai Cardiovascular (Other: Beijing Jiekai Cardiovascular Health Foundation)
Record Dates: First submitted 2025-03-14; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Mitral R; Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Structural Heart Surgery Assist System-assisted TEER. (Experimental)
  Interventions: Device: Structural Heart Surgery Assist System
- Manual TEER (e.g., MitraClip G4). (Placebo Comparator)
  Interventions: Device: Manual MitraClip G4

INTERVENTIONS:
Device: Structural Heart Surgery Assist System — Following femoral venous access and transseptal puncture, the steerable guide catheter and transcatheter mitral valve clip system are inserted and mounted onto the Structural Heart Surgery Assist System. The surgeon manipulates the joystick and controls on the operator console, guided by real-time animations on the human-machine interface that confirm the direction and range of device motion. Under fluoroscopic (DSA) and echocardiographic guidance, the system assists in performing edge-to-edge mitral valve repair. The procedure achieves regurgitation reduction by either creating a double-orifice configuration (A2/P2 segments) or approximating the opposing leaflets at the A1/P1 or A3/P3 regions.
  Arms: Structural Heart Surgery Assist System-assisted TEER.
Device: Manual MitraClip G4 — Manual MitraClip G4
  Arms: Manual TEER (e.g., MitraClip G4).

SUMMARY:
This trial aims to evaluate the safety and efficacy of the Structural Heart Surgery Assist System in assisting TEER for patients with moderate-to-severe or greater degenerative or functional mitral regurgitation (MR ≥3+). A prospective, multicenter, stratified randomized controlled design with non-inferiority comparison will be used. The experimental group will utilize the Structural Heart Surgery Assist System, while the control group will undergo manual TEER (e.g., MitraClip G4).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender.
2. Symptomatic moderate-to-severe or greater mitral regurgitation (MR ≥3+) confirmed by transthoracic and/or transesophageal echocardiography (TTE/TEE), with planned transcatheter edge-to-edge repair (TEER):

   For degenerative mitral regurgitation (DMR):

   -Deemed high-risk for surgical intervention by the heart team:STS score ≥8% for mitral valve replacement (MVR) mortality risk; ≥6% for mitral valve repair mortality risk; OR presence of ≥2 frailty indices (moderate-to-severe frailty); OR anatomical/technical barriers to surgery; OR ≥2 major organ dysfunctions unlikely to improve postoperatively; OR other high-risk factors per heart team assessment.OR patient declines surgery.

   For functional mitral regurgitation (FMR):
   * Persistent heart failure symptoms (NYHA Class III/IVa) despite guidelines directed medical therapy (GDMT), revascularization, or cardiac resynchronization therapy (CRT) for 1-3 months.
   * ≥1 hospitalization for heart failure within the past 12 months and/or BNP >150 pg/mL or NT-proBNP >600 pg/mL.
   * Left ventricular ejection fraction (LVEF) ≥20% and ≤50%, with left ventricular end-systolic diameter (LVESD) ≤70 mm.
3. Primary regurgitant jet is non-commissural and deemed treatable by the investigator (secondary jets, if present, must be clinically insignificant).
4. Volunteerly provides informed consent, understands the trial objectives, and agrees to comply with follow-up.

Exclusion Criteria:

1. Rheumatic mitral valve disease.
2. Uncorrected active infection.
3. Severe calcification or thickening in the clip coaptation zone, rendering TEER anatomically unsuitable.
4. Intracardiac mass, thrombus, or vegetation on echocardiography.
5. Severe right heart dysfunction (e.g., lower extremity edema with elevated jugular venous pressure and hepatomegaly) or severe pulmonary hypertension (echocardiographic systolic pulmonary artery pressure >70 mmHg).
6. Severe left heart dysfunction (LVEF <20%).
7. Acute myocardial infarction (AMI) within 30 days prior to the procedure.
8. Recent CABG, PCI, or TAVR within 30 days prior to the procedure.
9. Planned tricuspid/aortic valve or major vascular intervention within 30 days post-procedure.
10. Prior surgical or transcatheter mitral valve repair/replacement.
11. Thrombosis in access vessels (e.g., femoral vein, inferior vena cava) impeding catheter advancement.
12. Stroke/TIA within 30 days or severe carotid stenosis (>70% by ultrasound).
13. Cardiomyopathies or conditions including hypertrophic, restrictive, or infiltrative cardiomyopathy (e.g., amyloidosis, hemochromatosis, sarcoidosis), constrictive pericarditis, or active endocarditis.
14. Hemodynamic instability: Systolic blood pressure <90 mmHg without afterload-reducing agents, cardiogenic shock, requirement for intra-aortic balloon pump (IABP) or hemodynamic support.
15. Implanted pacemaker, CRT, or ICD within 30 days prior to the procedure.
16. End-stage heart failure (ACC/AHA Stage D), post-heart transplant, or listed for transplant.
17. Hypersensitivity or contraindications: ntolerance to anticoagulants, antiplatelet agents, or anesthesia, allergy to mitralclip materials (nickel/titanium, cobalt, chromium, polyester), severe contrast allergy precludes intervention.
18. Pregnant or breastfeeding.
19. Participation in other clinical trials (drug/device) without meeting primary endpoints.
20. Other contraindications per investigator judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2026-03-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
Surgical Success Rate | 7days
  All of the following conditions need to be met
  1. Successful implantation of 1 or more mitral clips (successful delivery and release of mitral clips with echocardiographic confirmation of leaflet clamping and successful withdrawal of the transcatheter mitral clip delivery system and manoeuvrable guide catheter);
  2. Transthoracic echocardiography showing a degree of mitral regurgitation ≤2+ (as evaluated by a third-party core laboratory) prior to discharge (up to 7 days).
  Calculation formula: Surgical success rate (%) = (number of cases achieving surgical success in each group/total number of cases in each group) × 100% for each group

SECONDARY OUTCOMES:
Instrumental technique success (trial group only) | Perioperative/Periprocedural
  Definition: Successful completion of transcatheter mitral valve edge-to-edge repair (TEER) using the Structural Heart Surgery Assist System without unplanned manual intervention.
  Unplanned Manual Intervention: Defined as conversion to manual operation during stages that the system is designed to assist (clip delivery and leaflet capture), per the Instructions for Use of the Structural Heart Surgery Assist System.
  Calculation formula: Instrumental technique success (%) = (number of cases achieving Instrumental technique success in trial group/total number of cases in trial group) × 100% for each group
Clinical Success Rate | 7days
  Criteria (all must be met):
  1. No intraoperative mortality related to the procedure.
  2. Successful delivery and deployment of the mitral valve clip, with retrieval of the transcatheter clip delivery system and steerable guide catheter.
  3. Placement of ≥1 mitral valve clip in the anatomically correct position.
  4. No unplanned surgeries or reinterventions related to the device or access site prior to discharge (within 7 days maximum).
  Calculation formula: Clinical Success Rate (%) = (number of cases achieving Clinical Success in each group/total number of cases in each group) × 100% for each group
Change in Mitral Regurgitation (MR) Severity | 7days/30days
  Assessed by comparing baseline Mitral Regurgitation (MR) Severity 7days and 30 days post-procedure.
  The severity of mitral regurgitation was classified as absent (0+), mild (1+), moderate (2+), moderately severe (3+), and severe (4+).
  Evaluation method: based on transthoracic echocardiography results.
Change in NYHA Functional Class | 30days
  Assessed by comparing baseline NYHA class to class at 30 days post-procedure.
Mitral Clip Implantation Time | Perioperative/Periprocedural
  Definition: Time from transseptal puncture initiation to successful withdrawal of the steerable guide catheter.
Fluoroscopy Time | Perioperative/Periprocedural
  Recorded using digital subtraction angiography (DSA) and defined as the cumulative X-ray exposure time from procedure start (defined as the first of: vascular access, anesthesia induction, or transesophageal echocardiography [TEE] probe insertion) to successful withdrawal of the steerable guide catheter.
Operator Radiation Exposure | Perioperative/Periprocedural
  Measured using radiation dosimeters worn by the operator, recording cumulative radiation dose from procedure start to guide catheter withdrawal

CONTACTS AND LOCATIONS:
Locations (1):
- Structural Heart Disease Unit, Xiamen Cardiovacular Hospital, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No